CLINICAL TRIAL: NCT03274557
Title: Treatment of Achilles Tendinose
Brief Title: Radiofrequence Microtenotomy for Treatment of Achilles Tendinose
Acronym: RFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/1277/REK sør-øst
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2017-09

CONDITIONS: Achilles Pain
Keywords: Achilles, tendinose, tendinopathy, pain
MeSH Terms: conditions — Tendinopathy; Pain

STUDY DESIGN:
Intervention Model Description: To evaluate improvement of VAS and functionality before and after treatment of Achilles tendinosis using radiofrequency-plasma based microtenotomy in comparison to traditional physical therapy.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency microtenotomy (Active Comparator): Treatment of Achilles tendinose with radio-frequency microtenotomy
  Interventions: Procedure: RFM
- Phusical therapy (Active Comparator): Supervised eccentric training
  Interventions: Procedure: RFM

INTERVENTIONS:
Procedure: RFM

SUMMARY:
Prospective randomized controlled study using radio-frequency microtenotomy or physical therapy (eccentric training) for treatment of Achilles tendinose

DETAILED DESCRIPTION:
Achilless tendinosis is a major clinical problem. There is a need for new studies to map the effectiveness of treatment. This study will compare treatment effectiveness between traditional physical therapy with surgical treatment using (RFM). The tendinosis grade will be evaluated using MRI and /or ultrasound before and after intervention. The outcome measurment include VAS and function using ( FAOS FOOT & ANKLE SURVEY) at 6,12 weeks and 6, 12 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain in Achilles tendon for at least 6 weeks.
* MR / ultrasound confirms diagnosis tendinose.
* Pain in sport and daily activities

Exclusion Criteria:

Other co-morbidity that constitutes contraindication for surgery, serious illness, bad compliance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 6.12 weeks and 6,12 months
  Pain reduction. Change of pain from baseline measured with VAS

SECONDARY OUTCOMES:
Function | 6.12 weeks and 6,12 months
  Change from baseline in functionality measured by (FAOS) FOOT & ANKLE SURVEY

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Al-Ani Z, Meknas D, Kartus JT, Lyngedal O, Meknas K. Radiofrequency Microtenotomy or Physical Therapy for Achilles Tendinopathy: Results of a Randomized Clinical Trial. Orthop J Sports Med. 2021 Dec 20;9(12):23259671211062555. doi: 10.1177/23259671211062555. eCollection 2021 Dec. PMID 34988234